CLINICAL TRIAL: NCT01822899
Title: DB2116134: A Randomized, Multi-center, Double-blind, Double-dummy, Parallel Group Study to Evaluate the Efficacy and Safety of Umeclidinium Bromide/Vilanterol Compared With Fluticasone Propionate/Salmeterol Over 12 Weeks in Subjects With COPD
Brief Title: A Study to Evaluate the Efficacy and Safety of Umeclidinium Bromide/Vilanterol Compared With Fluticasone Propionate/Salmeterol Over 12 Weeks in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116134
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Novel Dry Powder Inhaler (NDPI); umeclidinium bromide (UMEC); GSK573719; lung function; GW642444; salmeterol (SAL); fluticasone propionate (FP); vilanterol (VI); Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — vilanterol; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Umeclidinium bromide/Vilanterol + placebo ACCUHALER/DISKUS (Experimental): Subjects will receive UMEC/ VI 62.5/25 mcg, one inhalation administered once-daily in the morning via the NDPI and one placebo ACCUHALER/DISKUS administered as one inhalation each morning and evening.
  Interventions: Drug: Umeclidinium bromide/Vilanterol; Drug: Placebo ACCUHALER/DISKUS
- Fluticasone propionate/Salmeterol + placebo NDPI (Active Comparator): Subjects will receive FSC 500/50 mcg, administered as one inhalation each morning and evening via ACCUHALER/DISKUS + placebo administered once daily in the morning via NDPI.
  Interventions: Drug: Fluticasone propionate/Salmeterol; Drug: Placebo NDPI

INTERVENTIONS:
Drug: Umeclidinium bromide/Vilanterol — Dry white powder of UMEC 62.5 mcg per blister and VI 25 mcg per blister as NDPI with 30 doses (2 strips with 30 blisters per strip).
  Arms: Umeclidinium bromide/Vilanterol + placebo ACCUHALER/DISKUS
Drug: Placebo ACCUHALER/DISKUS — Dry white powder of matching placebo as multidose dry powder inhaler containing a foil strip with 60 blisters (1 strip with 60 blisters per strip).
  Arms: Umeclidinium bromide/Vilanterol + placebo ACCUHALER/DISKUS
Drug: Fluticasone propionate/Salmeterol — Dry white powder of fluticasone propionate 500 mcg per blister 50 mcg salmeterol per blister as multidose dry powder inhaler containing a foil strip with 60 blisters (1 strip with 60 blisters per strip).
  Arms: Fluticasone propionate/Salmeterol + placebo NDPI
Drug: Placebo NDPI — Dry white powder of matching placebo as NDPI with 30 doses (2 strips with 30 blisters per strip).
  Arms: Fluticasone propionate/Salmeterol + placebo NDPI

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, parallel group study. The purpose of this study is to compare the efficacy and safety of umeclidinium/vilanterol (UMEC/VI) and fluticasone propionate/salmeterol (FSC) in subjects with Chronic Obstructive Pulmonary Disease (COPD). Subjects who meet the eligibility criteria at Screening will complete a 7 to 14 day Run-in period. At the end of the run-in period, approximately 710 eligible subjects will be equally randomized (to complete at least 568 evaluable subjects) to one of the 2 treatment groups for 12 weeks: 1. UMEC/VI 62.5/25 micrograms (mcg) administered as one inhalation once-daily in the morning via the Novel dry powder inhaler (NDPI) + placebo administered as one inhalation each morning and evening via single multidose powdered inhaler (ACCUHALER/DISKUS) or 2. FSC 500/50 mcg administered as one inhalation each morning and evening via ACCUHALER/DISKUS + placebo administered once-daily in the morning via NDPI. A safety Follow-up assessment will be conducted approximately 7 days after the end of the study treatment (Early Withdrawal, if applicable). The total duration of subject participation will be approximately 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed Consent: A signed and dated written informed consent prior to study participation
* Age: Subjects 40 years of age or older at Visit 1
* Gender: Male or female subjects. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile); or Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the acceptable contraceptive methods listed in the protocol used consistently and correctly
* Diagnosis: established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society as follows: Chronic obstructive pulmonary disease is a preventable and treatable disease state characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.
* Smoking history: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day/20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar smoking cannot be used to calculate pack year history.
* Severity of disease: A pre and post-salbutamol FEV1/FVC ratio of <0.70 and a post-salbutamol FEV1 of >=30% and <=70% of predicted normal values calculated using NHANES III reference equations at Visit 1.
* Dyspnea: A score of >=2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Visit 1.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study
* Asthma: A current diagnosis of asthma
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject, who, in the opinion of the investigator, has any other significant respiratory condition in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Inactive tuberculosis in more than one lobe is exclusionary. Allergic rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, corticosteroid, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for pneumonia within 12 weeks prior to Visit 1
* History of COPD Exacerbation: A documented history of at least one COPD exacerbation in the 12 months prior to Visit 1 that required either oral corticosteroids, antibiotics, and/or hospitalization. Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Screening (Visit 1)
* 12-Lead ECG: An abnormal and significant electrocardiogram (ECG) finding from the 12-lead ECG conducted at Visit 1. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility.
* Medication Prior to Spirometry: Unable to withhold salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications Prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids - 12 weeks, Systemic, oral or parenteral corticosteroids - 6 weeks, Antibiotics (for lower respiratory tract infection) - 6 weeks, Cytochrome P450 3A4 strong inhibitors - 6 weeks, Herbal medications potentially containing oral or systemic steroids - 6 weeks, Inhaled corticosteroids (ICS) - 30 days, Long-acting beta2-agonist (LABA)/ICS combination products - 30 days, Phosphodiesterase 4 (PDE4) inhibitors (e.g., roflumilast) - 14 days, Inhaled long-acting anticholinergics - 7 days, Theophyllines - 48 hours, Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) - 48 hours, Oral beta2-agonists Long-acting-48 hours/Short-acting - 12 hours, Inhaled long acting beta2-agonists (LABA, e.g., salmeterol, formoterol, indacaterol) - 48 hours, Inhaled sodium cromoglycate or nedocromil sodium - 24 hours, Inhaled short acting beta2-agonists - 4 hours, Inhaled short-acting anticholinergics - 4 hours, Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products - 4 hours, Any other investigational medication - 30 days or within 5 drug half-lives (whichever is longer)
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator
* Inability to read: A subject will not be eligible for the study if in the opinion of the investigator the subject cannot read.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2013-04-04; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- Czechia (8):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Cvikov
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Kroměříž
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Třebíč
- Denmark (4):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Odense C
  - GSK Investigational Site, Roskilde
- Germany (9):
  - GSK Investigational Site, Dillingen an der Donau, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
- Hungary (12):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Farkasgyepű
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szikszó
- Netherlands (6):
  - GSK Investigational Site, Dordrecht
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Kloosterhaar
  - GSK Investigational Site, Sneek
- Poland (6):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Inowrocław
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Skierniewice
  - GSK Investigational Site, Słupsk
- Russia (15):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Kaluga
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Khantymansiysk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Petrozavodsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Pertersburg
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
- Spain (7):
  - GSK Investigational Site, Barcelona, Catalonia
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pama de Mallorca
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Singh D, Worsley S, Zhu CQ, Hardaker L, Church A. Umeclidinium/vilanterol versus fluticasone propionate/salmeterol in COPD: a randomised trial. BMC Pulm Med. 2015 Aug 19;15:91. doi: 10.1186/s12890-015-0092-1. PMID 26286141
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116134 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met the eligibility criteria at Screening (Visit 1) completed a 7- to 14-day Run-in Period, followed by a 12-week Treatment Period.
Pre-assignment Details: A total of 717 participants, representing the enrolled participants, were randomized to study treatment. Of these, 716 participants comprised the Intent-to-Treat Population (participants randomized to treatment who received >=1 dose of randomized study medication in the treatment period).
Groups:
- UMEC/VI 62.5/25 µg: Participants received umeclidinium bromide (UMEC) 62.5 micrograms (µg)/vilanterol (VI) 25 µg once daily (QD) each morning via a dry powder inhaler (DPI) and placebo twice daily (BID) (once in the morning and once in the evening) via a DPI for 12 weeks.
- FSC 500/50 µg: Participants received fluticasone propionate/salmeterol (FSC) 500 µg/50 µg BID (once in the morning and once in the evening) via a DPI and placebo administered QD via a DPI for 12 weeks.
Period: Overall Study
Arm/Group | UMEC/VI 62.5/25 µg | FSC 500/50 µg
Started | 358 | 358
Completed | 334 | 340
Not Completed | 24 | 18
Not completed — Adverse Event | 6 | 5
Not completed — Lack of Efficacy | 6 | 3
Not completed — Protocol Violation | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UMEC/VI 62.5/25 µg | FSC 500/50 µg | Total
Number analyzed (Participants) | 358 | 358 | 716
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (7.94) | 61.4 (8.06) | 61.6 (8.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 104 | 201
  Male | 261 | 254 | 515
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 358 | 358 | 716

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in 0 to 24 Hour Weighted Mean Serial Forced Expiratory Volume in One Second (FEV1) at Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 and post-dose FEV1 measurements at 5 and 15 minutes and 1, 3, 6, 9, 12 (pre-evening dose), 13, 15, 18, 23, and 24 hours after the morning dose. Analysis was performed using an analysis of covariance (ANCOVA) model with covariates of treatment, Baseline FEV1 (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), and smoking status.
Time Frame: Baseline and Day 84
Population: Intent-to-Treat (ITT) Population: all participants (par.) randomized to treatment who received at least one dose of randomized study drug in the Treatment Period. Par. analyzed were those with data available at the presented time point but all par. without missing covariate information and with >= post BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg | FSC 500/50 µg
Number analyzed (Participants) | 332 | 337
Liters | 0.166 (0.0122) | 0.087 (0.0121)
Statistical Analysis 1: Comparison: UMEC/VI 62.5/25 µg vs FSC 500/50 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 0.080, 95% CI 2-sided [0.046 to 0.113]

2. Secondary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) at Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. BL is defined as the mean of the assessments made 30 and 5 minutes (min) pre-dose on Treatment Day 1. Trough FEV1 on Day 85 is defined as the mean of the FEV1values obtained 23 and 24 hours after the previous morning's dosing (i.e., trough FEV1 on Day 85 is the mean of the FEV1 values obtained 23 and 24 hours after morning dosing on Day 84). Analysis was performed using a repeated measures model with covariates of treatment, BL (mean of the two assessments made 30 min and 5 min pre-dose on Day 1), smoking status, day, and day by BL and day by treatment interactions. The model used all available trough FEV1 values recorded on Days 28, 56, 84, and 85. Missing data were not directly imputed in this analysis; however, all non-missing data for a participant were used within the analysis to estimate the treatment effect for trough FEV1 at Day 85.
Time Frame: Baseline and Day 85
Population: ITT Population. Participants analyzed were those with data available at the presented time point; but, all participants without missing covariate information were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC/VI 62.5/25 µg | FSC 500/50 µg
Number analyzed (Participants) | 333 | 338
Liters | 0.151 (0.0126) | 0.062 (0.0125)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the follow-up contact (up to 13 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study drug in the Treatment Period.
Arm/Group | UMEC/VI 62.5/25 µg | FSC 500/50 µg
Serious Adverse Events (participants affected / at risk) | 7/358 | 2/358
Other Adverse Events (participants affected / at risk) | 39/358 | 32/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg (N=358) | FSC 500/50 µg (N=358)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC/VI 62.5/25 µg (N=358) | FSC 500/50 µg (N=358)
Headache (Nervous system disorders) | 33 | 25
Nasopharyngitis (Infections and infestations) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.